CLINICAL TRIAL: NCT06383884
Title: An Open Label, Phase 2 Basket Study of Patritumab Deruxtecan in Patients With Solid Tumor Harboring an NRG1 Fusion
Brief Title: Patritumab Deruxtecan in Patients With Solid Tumor Harboring an NRG1 Fusion
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Se-Hoon Lee, M.D. Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02-134
Record Dates: First submitted 2024-04-16; First posted 2024-04-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor, Adult
Keywords: Patritumab deruxtecan; NRG1 fusion
MeSH Terms: interventions — patritumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patritumab deruxtecan treatment arm (Experimental): Patritumab deruxtecan will be administered as an IV infusion Q3W on Day 1 of each 21-day cycle as a fixed dose regimen of 5.6 mg/kg Q3W.
  Interventions: Drug: Patritumab Deruxtecan

INTERVENTIONS:
Drug: Patritumab Deruxtecan — Patritumab deruxtecan will be administered as an IV infusion Q3W on Day 1 of each 21-day cycle as a fixed dose regimen of 5.6 mg/kg Q3W.
  Other Names: U3-1402

SUMMARY:
The NRG1 gene is located on chromosome 8 (8p12 region) and encode NRG1. NRG1 gene is translated to generate six different proteins (I-VI) and at least 31 isoforms. NRG1 proteins are structurally related to EGF and contain an EGF-like motif that binds and activates ErbB3 and ErbB4. Upon ligand binding, these receptors form homodimers or heterodimers, which results in phosphorylation of the intrinsic kinase domain, and activation of the PI3K-AKT, MAPK, and other pathways.

The overall incidence of NRG1 fusions is very rare. In many tumor types, only limited numbers of NRG1 fusion variant have been identified. By percentage, there is no organ dominance of the presence of NRG1 fusions. In an analysis of 21, 858 tumor specimens that underwent anchored multiplex PCR for targeted RNA sequencing, the prevalence of NRG1 fusions was 0.2%. Of these, CD74 was the most common partner (29%), followed by ATP1B1 (10%), SDC4 (7%), and RBPMS (5%), and most CD74-NRG1 fusions have been reported in patients with lung IMA. NRG1 fusions result in aberrant expression of the epidermal growth factor (EGF)-like domain of neuregulin-1 (NRG1) on the cell surface binds primarily to ErbB3 and ErbB4, leading to heterodimerization or oligomerization with other ERBB family members. NRG1-mediated activation of ErbB3 promotes dimerization with EGFR, ErbB2, and ErbB4. These partners phosphorylate ErbB3, forming docking sites for SH2-domain proteins, leading to pathologic activation of multiple signal transduction pathways, including the phosphoinositide 3-kinase (PI3K) pathway. Subsequently, ErbB3 expression was noted at high levels, and the proteins were phosphorylated, in fusion-positive cases. Targeting ErbB3 signaling therefore represents a promising therapeutic approach for patients with NRG1 fusion-positive malignancies.

DETAILED DESCRIPTION:
This is a global, multicenter, open-label, Phase 2 study exploring the efficacy and safety of patritumab deruxtecan in patients with NRG1 fusion solid tumor. Patients with tumor harboring NRG1 fusion will be identified through previously documented mutation testing performed prior to screening. The presence of NRG1 fusion will be retrospectively confirmed by central testing via next generation sequencing (NGS) or FISH or Anchored multiplex PCR for targeted RNA sequencing (AMP). The study has a basket design and includes several cohorts, either defined by an actionable somatic mutation and tumor histology.

Patritumab deruxtecan will be dosed at 5.6mg/kg as an itravenous (IV) infusion administered on Day 1 of each 21-day cycle. Dose reductions or interruptions, and initiation of supportive care, are allowed as deemed appropriate by the investigator.

The study start date is the date when the first subject has signed the main informed consent. A subject is eligible to be enrolled into the interventional phase of the study when the Investigator or designee has obtained written consent, has confirmed all eligibility criteria have been met by the subject, and all Screening procedures have been completed.

A Simon's optimal 2-stage design (with significance level 5%, power of 80%) will be used to determine whether patritumab deruxtecan has sufficient activity to warrant further development. The null hypothesis is carried through into the second stage before it is rejected or not. Early study termination will be permitted if data at the first stage indicate that the treatment is ineffective.

As the range of ORR in NRG1 fusion patients treated with chemotherapy or chemoimmunotherapy was found to be 0% to 13%, the investigators considered the average 6% will be considered unacceptable, whereas the ORR of patients who treated with afatinib was 25%, the investigators hypothesized the average of ORR 25% will merit further study (alternative hypothesis).

In the first stage, enrollment will continue until 7 patients received at least one dose of study treatment and completed the first tumor assessment by the investigator (response evaluable). If no responses are observed, the second stage for the cohort must be discontinued. Otherwise, 23 additional response evaluable patients will be accrued for a total of 30 patients in the cohort, considering 15% of dropout rate. The null hypothesis will be rejected if at least 4 responses are observed in Stage 2.

The study will be divided into 3 periods: a Screening Period, Treatment Period, and Follow-up Period.

The primary analysis of ORR will be conducted after all enrolled subjects have either a minimum of 9 months of follow-up or have discontinued from the study earlier. The final analysis will occur after all subjects have discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Sign and date the tissue informed consent form (ICF) and the main ICF, prior to the start of any study-specific qualification procedures.
* Male or female participants aged ≥18 years (follow local regulatory requirements if the legal age of consent for study participation is >18 years old).
* Histologically or cytologically documented locally advanced or metastatic solid tumor not amenable to curative surgery or radiation.
* Documentation of NRG1 fusion detected from tumor tissue or blood sample, including but not limited to TruSightOncology-500, Guardant-360 or FoundationOne®CDx (F1CDx).
* At least 1 measurable lesion confirmed by investigator as per RECIST v1.1
* At least 1 measurable lesion confirmed per RECIST v1.1
* Consented and willing to provide required tumor tissue of sufficient quantity (as defined in the Laboratory Manual) and of adequate tumor tissue content (as confirmed by hematoxylin and eosin [H&E] staining). Required tumor tissue can be provided as either:

  1. Pretreatment tumor biopsy from at least 1 lesion not previously irradiated and amenable to core biopsy OR
  2. Archival tumor tissue collected from a biopsy performed within 3 months prior to signing of the tissue consent and since progression while on or after treatment with the most recent cancer therapy regimen.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1 at Screening.
* Has adequate bone marrow reserve and organ function based on local laboratory data within 14 days prior to Cycle 1 Day

  1. Platelet count: ≥100,000/mm^3 or ≥100 × 10^9/L (platelet transfusions are not allowed up to 14 days prior to Cycle 1 Day 1 to meet eligibility)
  2. Hemoglobin: ≥9.0 g/dL (transfusion and/or growth factor support is allowed)
  3. Absolute neutrophil count: ≥1500/mm^3 or ≥1.5 × 10^9/L
  4. Serum creatinine (SCr) or creatinine clearance (CrCl): SCr ≤1.5 × upper limit of normal (ULN), OR CrCl ≥30 mL/min as calculated using the Cockcroft-Gault equation or measured CrCl
  5. Aspartate aminotransferase/alanine aminotransferase: ≤3 × ULN (if liver metastases are present, ≤5 × ULN)
  6. Total bilirubin: ≤1.5 × ULN if no liver metastases (<3 × ULN in the presence of documented Gilbert's syndrome [unconjugated hyperbilirubinemia] or liver metastases)
  7. Serum albumin: ≥2.5 g/dL
  8. Prothrombin time (PT) or PT-International normalized ratio (INR) and activated partial thromboplastin time (aPTT)/PTT: ≤1.5 × ULN, except for subjects on coumarin-derivative anticoagulants or other similar anticoagulant therapy, who must have PT-INR within therapeutic range as deemed appropriate by the Investigator

Exclusion Criteria:

* Any history of interstitial lung disease (including pulmonary fibrosis or radiation pneumonitis) has current interstitial lung disease (ILD) or is suspected to have such disease by imaging during screening.
* Clinically severe respiratory compromise (based on Investigator's assessment) resulting from intercurrent pulmonary illnesses including, but not limited to:

  1. Any underlying pulmonary disorder (eg, pulmonary emboli within 3 months prior to the study enrollment, severe asthma, severe chronic obstructive pulmonary disease [COPD]), restrictive lung disease, pleural effusion);
  2. Any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (eg, rheumatoid arthritis, Sjogren's syndrome, sarcoidosis); OR prior complete pneumonectomy.
* Is receiving chronic systemic corticosteroids dosed at >10 mg prednisone or equivalent anti-inflammatory or any form of immunosuppressive therapy prior to enrollment. Participants who require use of bronchodilators, inhaled or topical steroids, or local steroid injections may be included in the study.
* Evidence of any leptomeningeal disease.
* Evidence of clinically active spinal cord compression or brain metastases.
* Inadequate washout period prior to Cycle 1 Day 1, defined as:

  1. Whole brain radiation therapy <14 days or stereotactic brain radiation therapy <7 days;
  2. Any cytotoxic chemotherapy, investigational agent or other anticancer drug(s) from a previous cancer treatment regimen or clinical study (other than EGFR TKI), <14 days or 5 half-lives, whichever is longer;
  3. Monoclonal antibodies, other than immune checkpoint inhibitors, such as bevacizumab (anti-VEGF) and cetuximab (anti-EGFR) <28 days;
  4. Immune checkpoint inhibitor therapy <21 days;
  5. Major surgery (excluding placement of vascular access) <28 days;
  6. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation <28 days or palliative radiation therapy <14 days; or
  7. Chloroquine or hydroxychloroquine <14 days.
* Prior treatment with an anti-human epidermal growth factor receptor 3 (HER3) antibody or single-agent topoisomerase I inhibitor.
* Prior treatment with an antibody drug conjugate (ADC) that consists of any topoisomerase I inhibitor
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0, Grade ≤1 or baseline. Participants with chronic Grade 2 toxicities may be eligible at the discretion of the Investigator.
* Has history of other active malignancy within 3 years prior to enrollment, except:

  1. Adequately treated non-melanoma skin cancer;
  2. Superficial bladder tumors (Ta, Tis, T1);
  3. Well-differentiated thyroid cancer
  4. Adequately treated intraepithelial carcinoma of the cervix uteri;
  5. Low risk non-metastatic prostate cancer (with Gleason score <7, and following local treatment or ongoing active surveillance);
  6. Any other curatively treated in situ disease.
* Uncontrolled or significant cardiovascular disease prior to Cycle 1 Day 1
* Active hepatitis B and/or hepatitis C infection, such as those with serologic evidence of viral infection within 28 days of Cycle 1 Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 12 month after completion of enrollment
  assessed by investigator per RECIST v1.1

SECONDARY OUTCOMES:
Duration of response (DoR) | up to 30 month
  DoR as assessed by investigator per RECIST v1.1
Progression-free survival(PFS) | up to 30 month
  PFS as assessed by investigator per RECIST v1.1
Disease-control rate(DCR) | up to 30 month
  DCR as assessed by investigator and Investigator per RECIST v1.1
Best percentage change in the SoD of measurable tumors | up to 30 month
  SoD as assessed by investigator per RECIST V1.1
Overall survival(OS) | up to 30 month
  Death date is collected until the subject discontinues the study.

OTHER OUTCOMES:
Incidence of Adverse events (CTCAE v5.0) | From the start to the end of the subject's study, an average of 6 month
  Safety during the study

CONTACTS AND LOCATIONS:
Overall Officials: Se-Hoon Lee, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No